CLINICAL TRIAL: NCT06353867
Title: The Effect of Group Exercise on Balance and Attention Level in Children With Special Needs
Brief Title: The Effect of Group Exercise in Children With Special Needs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Gedik University (Other)
Responsible Party: Principal Investigator, Gokce Kartal, MSc,PT, Istanbul Gedik University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 56365223-050.01.04-2023.13754
Record Dates: First submitted 2024-04-03; First posted 2024-04-09 (Actual); Last update posted 2024-04-09 (Actual); Status verified 2024-04

CONDITIONS: Developmental Disability; Child Autism
Keywords: developmental disability; balance; attention; group exercise
MeSH Terms: conditions — Developmental Disabilities; Autistic Disorder

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Group Exercise (Experimental)
  Interventions: Other: Group Exercise

INTERVENTIONS:
Other: Group Exercise — The children with special needs included in the study were included in group exercises for 45 minutes 2 days a week in groups of 10 children each. Group exercises were planned as balance and coordination exercises including warm-up and cool-down periods. In the warm-up and cool-down periods, counting in place and balance exercises were performed. The exercises included tasks such as side walking, tandem walking, walking on a balance board, walking in a figure 8, walking over obstacles, throwing a ball to the person next to him/her while passing through cones, and throwing a ball by jumping while passing through cones.The exercises were made more difficult by following a progressive method every 2 weeks. The exercises were performed in 3 sets of 5 repetitions under the supervision of a physiotherapist.

SUMMARY:
Thirty children with special needs were included in the study. Participants engaged in group exercises twice a week for four weeks, including warm-up and cool-down periods, with the goal of improving balance. The participants' balance was assessed using the Bruininks-Oseretsky Motor Proficiency Test Short Form (Balance Parameters), Pediatric Balance Scale; functional mobility was evaluated using the Timed Up and Go Test, and attention level was assessed using the Stroop Test before and after the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 6-15 years with special needs
* Able to walk independently

Exclusion Criteria:

* Children with visual problems,
* Any orthopaedic, rheumatic or neurological problems affecting balance,
* Any contraindication to exercise

Ages: 6 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2022-12-27 (Actual); Primary Completion 2023-04-15 (Actual); Study Completion 2023-04-25 (Actual)

PRIMARY OUTCOMES:
Bruininks-Oseretsky Motor Competence Test Short Form Balance Subtest (Balance Subtest of BOT 2-KF) | Baseline and after the interventions (4th week)
  1. Standing on the dominant leg on the balance board: The participant will be asked to stand on the balance board with his/her eyes open on his/her dominant foot, looking at the target, with his/her hands on his/her waist and the other leg parallel to the ground for 10 seconds. Scoring will be recorded as 0-0.9 s 0 points, 1-2.9 s 1 point, 3-5.9 s 2 points, 6-9.9 s 3 points and 10 s 4 points according to the duration of standing on one leg.
  2. Tandem (heel-thumb) walking on the walking line: The participant will be asked to place his/her hands on his/her waist and walk along the walking line. When 6 steps are completed, the test is stopped. Steps that does not go beyond the line are evaluated. Scoring is done as 0 step 0 points, 1-2 steps 1 point, 3-4 steps 2 points, 5 steps 3 points and 6 steps 4 points.
Paediatric Balance Scale | Baseline and after the interventions (4th week)
  The version consisting of 14 sections and each section scored between 0-4 is used to evaluate the balance status of the participants.
Functional Reach Test | Baseline and after the interventions (4th week)
  The participant is asked to reach as far as he/she can horizontally at the level of a tape measure fixed to the wall with arms at 90 flexion. The test is repeated 3 times and the measurements are averaged.
Timed Up and Go Test | Baseline and after the interventions (4th week)
  It will be applied to assess balance and functional ambulation. The participant is asked to get up from a chair, walk 3 metres, turn around and sit down again. The time it took to complete the test will be recorded.
Stroop Test | Baseline and after the interventions (4th week)
  The Stroop Test is among the neuropsychological tests frequently used to assess attention level and executive functions in children. Participants' time to complete the test is recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Gokce Kartal, PT, Principal Investigator — Marmara University
Locations (1):
- Marmara University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No